CLINICAL TRIAL: NCT02800278
Title: Characteristics and Outcomes of Odontoid Fragility Fractures in Elderly
Acronym: FOOP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: CHU de Nice RHUM
Record Dates: First submitted 2016-05-18; First posted 2016-06-15 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Odontoid Fracture; Osteoporosis; Surgery
MeSH Terms: conditions — Osteoporosis | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: observational — describe bone status and outcome of odontoid fracture

SUMMARY:
Usually, cervical spine fractures are not considered as osteoporotic fractures. However, recent studies show that odontoid fractures are the most common fractures of the cervical spine in elderly and may occur in a context of low trauma energy. Thus, the goal of this observationnal study is :

* to describe the different type of odontoid fracture and to characterize bone status in elderly patient (>65 y) who underwent odontoid fracture in a context of low trauma energy.
* To describe short and long term outcomes

DETAILED DESCRIPTION:
All patients over 65 y admitted for low trauma odontoid fracture will be consecutively included in the study after informed consent. The investigators will record:

* clinical risk factor of osteoporosis and health habits including accomodation
* type of fracture and characterization of the odontoid fracture on imaging (standard X ray / MRI / QCT)
* Bone status : bone mineral density on DXA, lab tests for secondary osteoporosis check-up, previous vertebral fracture on VFA or X ray
* osteoporosis managment : nutrition, vitamin D, anti-osteoporotic drugs
* treatment of the fracture : surgical / non surgical
* adverse event during hospitalization
* lenght of hospital stay
* type of discharge

Follow-up à 3 and 12 months : dead vs alive ; accomodation ; autonomy ; new fracture

ELIGIBILITY:
Inclusion Criteria:

* all patients over 65 y admitted for low traumat odontoid fracture

Exclusion Criteria:

* patient < 65 y
* traumatic odontoid fracture

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: all patients over 65 y admitted for low traumat odontoid fracture
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
bone status at the time of odontoid fracture: bone mineral density, prevalent osteoporotic fracture, vitamin D status | from date of inclusion until to 3 weeks after the event. Inclusion will be proposed within 2 weeks after the fracture
  clinical risk factor of osteoporosis, prevalent clinical osteoporotic fracture, bone mineral density measured by DXA, vertebral fracture assessment to detect other vertebral fracture, serum concentration in 25OHvitamin D

SECONDARY OUTCOMES:
mortality | during hospitalization - 3 and 12 months after inclusion
  mortality after odontoid fracture during hospitalization and at 3 and 12 monts
morbidity | during hospitalization - 3 and 12 months after inclusion
  incident osteoporotic fracture, adverse event such as infection, cardiovascular event, neurological event
loss of autonomy | discharge, 3 and 12 months
  lenght of hospital stay, type of discharge (home, nursing home, rehabilitation bed care, institutionalized accomodation

CONTACTS AND LOCATIONS:
Overall Officials: veronique breuil, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU, Nice, France

IPD SHARING:
Plan to Share IPD: No